CLINICAL TRIAL: NCT00866684
Title: Prevention of Skin Cancer in High Risk Patients After Conversion to a Sirolimus-based Immunosuppressive Protocol
Acronym: PROSKIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient patient recruitment
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Petra Reinke, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROSKIN 01
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Skin Cancer
Keywords: Renal transplant-patients with high-risk for skin cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — Sirolimus; Azathioprine; Mycophenolic Acid; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Sirolimus (Experimental): Patients will receive Sirolimus in addition to their previous immunosuppressive therapy.
  Interventions: Drug: Sirolimus
- 2 Standard (Active Comparator): Patients will stay on their previous immunosuppressive regimen.
  Interventions: Drug: Azathioprine; Drug: Mycophenolate; Drug: Ciclosporin; Drug: Tacrolimus

INTERVENTIONS:
Drug: Sirolimus — Treatment arm Dosage: 4-8 micrograms/litre; Route of administration: oral use; Frequency: one tablet per day
  Other Names: Rapamune, ATC code: L04AA10
  Arms: 1 Sirolimus
Drug: Azathioprine — control arm Dosage form: Coated tablet; dosage: 1-4 milligrams/kilogram; Frequency: daily; Duration: 24 month
  Other Names: ATC code: L04AX01
  Arms: 2 Standard
Drug: Mycophenolate — Control arm Dosage form: Tablet; dosage: 2 gram; Frequency: daily; Duration: 24 month
  Other Names: ATC code: L04AA06
  Arms: 2 Standard
Drug: Ciclosporin — Control arm Dosage form: Capsule; Dosage: 50-80 micrograms/litre; Frequency: daily; Duration: 24 month
  Other Names: ATC code: L04AA01
  Arms: 2 Standard
Drug: Tacrolimus — Control arm Dosage form: Capsule; dosage: 3-5 micrograms/litre; Frequency: daily; Duration: 24 month
  Other Names: ATC code: L04AA05
  Arms: 2 Standard

SUMMARY:
Transplant recipients have a high risk to develop skin malignancies. This effect depends on the one hand on the immunosuppressive drugs themselves (i.e., azathioprine) and relates on the other hand on the dosage (i.e., calcineurin-inhibitors). Based on the encouraging results of previous, retrospective studies on patients treated with Sirolimus (SRL), these patients should be switched to an immunosuppressive regime including SRL, decreasing the dosage of calcineurin-inhibitors or converting from former immunosuppression. A conversion to a SRL-based therapy is effective in immunosuppression and safe regarding graft and patient survival.

This study was designed to assess whether a switch to a SRL-immunosuppressive therapy decreases the incidence/reoccurrence of skin neoplasm.

DETAILED DESCRIPTION:
Patients who meet all inclusion criteria will be included into the study and randomised. If converted to SRL, patients will take SRL according to the investigator's instructions and medication label, once daily preferably 4 hours after calcineurin-inhibitor medication or in case without calcineurin-inhibitor co-medication in the morning. The dose of SRL will be correlated to the former immunosuppressive therapy according to the study's conversion protocol.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of renal allograft with current actinic keratosis I or II or successfully treated actinic keratosis III (inclusion possible immediately after completed wound healing from surgical excision), invasive squamous cell carcinoma (SCC), basal cell carcinoma and/or premalignant neoplastic skin lesions
* Age 18 years and older
* Minimum period of 6 month after renal transplantation
* Stable renal function and a calculated creatinine clearance of at least 40 ml/min
* Written informed consent
* Proteinuria ≤ 800 mg/d at time of enrolment
* Successfully treated solid tumor (no recurrence or metastasis in the last 2 years)

Exclusion Criteria:

* Current Sirolimus- or Everolimus- intake
* Instable graft function (creatinine clearance < 40 ml/min)
* Graft rejection within the 3 previous months
* Proteinuria > 800 mg/d
* Non-controlled hyperlipidemia (Cholesterol >7,8 mmol/l, Triglycerides > 4)
* Leucopenia < 2500/nl
* Thrombocytopenia < 90/nl
* Pregnancy or breastfeeding
* Women of childbearing age without highly effective contraception (= defined as those which result in a low failure rate (i.e. less than 1 % per year))
* Known allergy to macrolides
* Current participation in other studies
* Refusal to sign informed consent form
* Neoplasm other than defined as inclusion criteria
* All contraindications to SRL (see package insert, appendix)
* Persons who are detained officially or legally to an official institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2011-04-19 (Actual); Study Completion 2011-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petra Reinke, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (15):
- Germany (15):
  - Universitätsklinikum Erlangen, Hautklinik, Erlangen, Bavaria
  - Universitätsklinikum Erlangen, Medizinische Klinik IV, Erlangen, Bavaria
  - Klinikum der LMU München, Medizinische Poliklinik Innenstadt, München, Bavaria
  - Klinikum der LMU München, Klinik und Poliklinik für Dermatologie, München, Bavaria
  - Klinikum rechts der Isar, Klinik und Poliklinik für Dermatologie und Allergologie, München, Bavaria
  - Klinikum rechts der Isar, II. Medizinische Klinik und Poliklinik, München, Bavaria
  - Universität Regensburg, Dermatologie, Regensburg, Bavaria
  - Universität Regensburg, Nephrologie Innere Medizin II, Regensburg, Bavaria
  - Kliniken der Stadt Köln, Medizinische Klinik I, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Münster, Klinik und Poliklinik für Hautkrankheiten, Münster, North Rhine-Westphalia
  - Universitätsklinikum Münster, Med. Klinik und Poliklinik D, Münster, North Rhine-Westphalia
  - HELIOS Klinikum Wuppertal, Zentrum für Dermatologie, Allergologie und Umweltmedizin, Wuppertal, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Klinik für Dermatologie, Venerologie und Allergologie, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein, Klinik für Nieren- und Hochdruckkrankheiten, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin, Klinik für Dermatologie, Venerologie und Allergologie, Berlin

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Sirolimus: Patients will receive Sirolimus in addition to their previous immunosuppressive therapy.
  Sirolimus: Treatment arm Dosage:
  adapted to serum level: 4-8 micrograms/litre; Route of administration: oral use; Frequency: once per day (Tablets)
- 2 Standard: Patients will stay on their previous immunosuppressive regimen.
  Azathioprine: control arm Dosage form: Coated tablet; dosage: 1-4 milligrams/kilogram; Frequency: daily; Duration: 24 month
  Mycophenolate: Control arm Dosage form: Tablet; dosage: 2 gram; Frequency: daily; Duration: 24 month
  Ciclosporin: Control arm Dosage form: Capsule; Dosage adapted to serum level: 50-80 micrograms/litre; Frequency: daily; Duration: 24 month
  Tacrolimus: Control arm Dosage form: Capsule; dosage adapted to serum level: 3-5 micrograms/litre; Frequency: daily; Duration: 24 month
Period: Overall Study
Arm/Group | 1 Sirolimus | 2 Standard
Started | 25 | 19
Completed | 25 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Sirolimus: Patients will receive Sirolimus in addition to their previous immunosuppressive therapy.
  Sirolimus: Treatment arm Dosage adapted to serum level: 4-8 micrograms/litre; Route of administration: oral use; Frequency: once per day (Tablets)
- Total: Total of all reporting groups
Arm/Group | 1 Sirolimus | 2 Standard | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 9 | 26
  >=65 years | 8 | 10 | 18
Age, Continuous [Median (Full Range); unit: years] | 64.4 [18 to 75] | 59.6 [18 to 75] | 61.68 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 18 | 13 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Events of Reoccurrence of Skin Cancer
Description: Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Time Frame: 24 month
Measure: Number; unit: Event
Arm/Group | 1 Sirolimus | 2 Standard
Number analyzed (Participants) | 25 | 19
Event | 25 | 19

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- 1 Sirolimus: Patients will receive Sirolimus in addition to their previous immunosuppressive therapy.
  Sirolimus: Treatment arm Dosage adapted to Serum level: 4-8 micrograms/litre; Route of administration: oral use; Frequency: once per day (tablet)
- 2 Standard: Patients will stay on their previous immunosuppressive regimen.
  Azathioprine: control arm Dosage form: Coated tablet; dosage: 1-4 milligrams/kilogram; Frequency: daily; Duration: 24 month
  Mycophenolate: Control arm Dosage form: Tablet; dosage: 2 gram; Frequency: daily; Duration: 24 month
  Ciclosporin: Control arm Dosage form: Capsule; Dosage adapted to Serum level 50-80 micrograms/litre; Frequency: daily; Duration: 24 month
  Tacrolimus: Control arm Dosage form: Capsule; dosage adapted to Serum level 3-5 micrograms/litre; Frequency: daily; Duration: 24 month
Arm/Group | 1 Sirolimus | 2 Standard
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/19
Serious Adverse Events (participants affected / at risk) | 15/25 | 7/19
Other Adverse Events (participants affected / at risk) | 19/25 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Sirolimus (N=25) | 2 Standard (N=19)
Multiple squamous cell carcinomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (25) | 7 (14)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Sirolimus (N=25) | 2 Standard (N=19)
Urinary tract infection (Renal and urinary disorders) | 19 (60) | 9 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes